CLINICAL TRIAL: NCT00616213
Title: A Phase I, Multi-Center, Open-Label, Dose Escalation Trial of the Safety and Pharmacokinetics of Intravenous PR104 Given With Prophylactic G-CSF in Subjects With Solid Tumors
Brief Title: PR104 and G-CSF in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Proacta, Incorporated (Industry)
Responsible Party: Brenda Gibson, Assoc. Director, Proacta, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR104-1004; PROACTA-PR-104-1004
Record Dates: First submitted 2008-02-14; First posted 2008-02-15 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; PR-104; fluoromisonidazole

INTERVENTIONS:
Biological: filgrastim — filgrastim will be administered at a standard dose and schedule
  Other Names: Neupogen; G-CSF
Drug: PR104 — PR104 is administered intravenously once every 21 days
  Other Names: PR-104
Other: F-18-fluoromisonidazole — F-18-fluoromisonidazole is administered intravenously prior to performance of PET scan
  Other Names: FMISO

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as PR-104, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Colony-stimulating factors, such as G-CSF, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Giving PR-104 together with G-CSF may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of PR-104 when given together with G-CSF in treating patients with solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of PR-104 in combination with filgrastim (G-CSF) in patients with solid tumors.

Secondary

* Characterize the safety of this regimen in these patients.
* Evaluate the pharmacokinetics of PR-104 and its alcohol metabolite.
* Evaluate the rate of hypoxia in various solid tumors using F-MISO PET (18F-fluoromisonidazole positron emission tomography) imaging.
* Assess for antitumor toxicity in these patients.
* Collect plasma samples for the assessment of potential biomarkers of tumor hypoxia.

OUTLINE: This is a multicenter, dose-escalation study of PR-104.

Patients receive PR-104 IV over 1 hour on day 1 and filgrastim (G-CSF) on day 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo 18F-fluoromisonidazole PET scans at baseline and prior to course 3 to assess tumor hypoxia.

Patients undergo blood sample collection periodically during course 1. Samples are analyzed for the pharmacokinetics of PR-104 and for identification of biomarkers for tumor hypoxia.

After completion of study treatment, patients are followed at 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumors
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-1
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Hemoglobin ≥ 9 g/dL (no red blood cell transfusions allowed)
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* PTT ≤ 1.5 times normal
* Serum creatinine ≤ 1.5 times ULN
* ALT or AST ≤ 2 times ULN (≤ 5 times ULN if liver metastases are present)
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 30 days after completion of study therapy
* Able to read, understand, and provide written informed consent

Exclusion criteria:

* Evidence of a significant medical disorder or laboratory finding that, in the opinion of the investigator, compromises the patient's safety during study participation, including any of the following:

  * Uncontrolled infection or infection requiring a concomitant parenteral antibiotic
  * Uncontrolled diabetes
  * Congestive heart failure
  * Myocardial infarction within the past 6 months
  * Chronic renal disease
  * Coagulopathy (excluding prophylactic anticoagulation)
* Known HIV positivity
* Hepatitis B sAg-positive or known to be hepatitis C-positive with abnormal liver function tests

PRIOR CONCURRENT THERAPY:

* No more than 3 prior myelosuppressive chemotherapy regimens

  * Patients who have received more than 3 prior myelosuppressive regimens may be eligible, if considered to have adequate marrow, based on prior exposure to 1 of the following regimens:

    * Minimally myelosuppressive regimens
    * Limited courses of myelosuppressive regimens
* More than 4 weeks since prior and no other concurrent licensed or investigational anticancer treatment (6 weeks for nitrosoureas or mitomycin C)
* More than 24 hours since any prior radiotherapy and no likelihood of toxicity from this therapy
* More than 4 weeks since major surgery
* No prior radiotherapy to > 20% of bone marrow
* No prior high-dose chemotherapy (including either myeloablative or non-myeloablative transplantations)
* Prior and concurrent androgen deprivation therapy allowed
* Concurrent systemic steroids allowed, provided the patient has been on a stable dose for at least 2 weeks prior to first dose of PR-104
* No concurrent irradiation therapy (palliative or therapeutic), unless given in the absence of tumor progression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of PR-104 | 3 weeks (cycle 1)

SECONDARY OUTCOMES:
Safety profile using CTCAE v3 criteria
Dose-limiting toxicity of PR-104
Pharmacokinetics of PR-104 and its alcohol metabolite in blood
Anti-tumor activity
Biomarkers of tumor hypoxia

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Virginia G. Piper Cancer Center at Scottsdale Healthcare - Shea, Scottsdale, Arizona
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- Waikato Hospital, Hamilton, New Zealand